CLINICAL TRIAL: NCT03658915
Title: Validity and Reliability of Smartphone Use in Measuring Joint Position Sense in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Aliaa Rehan Youssef (Other)
Responsible Party: Sponsor-Investigator, Aliaa Rehan Youssef, Principle investigator, Cairo University
Organization: Cairo University (Other)
Other Study IDs: AY32
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Knee Osteoarthritis
Keywords: Position sense; Smartphone; Validity; Reliability; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoarthritis: Thirty symptomatic knee with osteoarthritis will be recruited according to the following criteria:
  INCLUSION CRITERIA:
  1. Referred with a confirmed diagnosis of unilateral or bilateral OA of the knee based on the following criteria.
     1.1. Morning stiffness < 30 minutes, 1.2. Crepitus on active knee movement. 1.3. Bony enlargement either palpable or visible in radiographs. 1.4. Bony tenderness.
  2. Age 40-60 years old.
  EXCLUSION CRITERIA:
  1. Steroid injection within the past 2 months.
  2. Presence of neurologic disorders.
  3. Presence of of orthopedic diseases or trauma in the lower extremity or spine within the past year.
  6. Severe pain with active movement 7. Poor memory or cognitive function
  Interventions: Device: Smartphone application (Goniometer Pro )
- Control: Thirty asymptomatic knee will be recruited for this study. Control group participants will be age-matched to the osteoarthritis group, and should have no pain or other relevant clinical symptoms in lower quadrant.
  Interventions: Device: Smartphone application (Goniometer Pro )

INTERVENTIONS:
Device: Smartphone application (Goniometer Pro ) — Knee repositioning error will be measured simultaneously by smartphone and Biodex isokinetic dynamometer by a single blind assessor. All assessments will be done with eyes closed and repeated over two separate sessions, with one-week interval in-between. For active repositioning, the participant will actively extend the knee to reach a predetermined target position45° flexion at an angular velocity of 10°/sec. For passive knee repositioning, the isokinetic dynamometer will move the knee at 5°/s to a predetermined angle between 5° and 80° of flexion and the participant should stop the movement when the predetermined angle is reached.

SUMMARY:
This study will investigate the concurrent validity and intra-rater reliability of using smartphone in assessing joint position sense in patient with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is the most common arthritis. Such disease is complicated by many musculoskeletal dysfunction such as disturbed joint position sense, which impairs their ability to perform their regular daily activities. As rehabilitation should target impairment in function, it is essential that therapists assess joint sense during baseline and follow-up evaluation of patients to decide on needed therapeutic interventions. Joint position sense can be assessed by various methods such as motion tracking systems and the isokinetic dynamometer, yet these equipment are expensive and are not readily available at regular clinical settings.

Smartphone has been introduced as an assessment tool in rehabilitation of musculoskeletal disorders. For the knee joint, smartphone has been validated for measuring range of motion and joint position sense in healthy population, yet it has never been validated in patients with knee osteoarthritis. Therefore, this study will investigate smartphone validity and reliability as an assessment tool of knee position sense in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be referred to the outpatient clinic of the faculty of Physical Therapy and Medicine, Cairo University with a confirmed diagnosis of unilateral or bilateral osteoarthritis of the knee and having one or more of the following criteria (ASo, 2000).
* Morning stiffness for less than 30 minutes.
* Crepitus on active knee movement.
* Bony enlargement either palpable or visible in radiographs.
* Bony tenderness at joint margins.
* Age 40-60 years old.

Exclusion Criteria:

* Steroid injection within 2 months prior to inclusion.
* Presence of neurologic disorders (e.g., stroke, Parkinson's disease, or poliomyelitis). •Presence of other rheumatoid or orthopedic disorders in the lower extremity or spine. •A recent history of a lower extremity fracture with in the past year.
* History of ligament deficiency, such as anterior cruciate ligament or meniscal injury.
* Severe pain with active movement.
* Poor memory or cognitive function.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects between 40 to 60 years old with symptomatic knee osteoarthritis and age-matched healthy control.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
concurrent validity of smartphone against isokinetic dynamometry in measuring joint position sense. | One day
  The extent to which a measure by Goniometer Pro application related to an outcome which is joint position sense in isokinetic dynamometer

SECONDARY OUTCOMES:
Intrarater reliability of smartphone measurements | 1 week
  same investigator will repeat joint position sens assessment using smartphone application

CONTACTS AND LOCATIONS:
Overall Officials: Aliaa Rehan Youssef, PhD, Principal Investigator — Cairo University, Faculty of Physical Therapy
Locations (1):
- Faculty of Physical Therapy, Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Background] Recommendations for the medical management of osteoarthritis of the hip and knee: 2000 update. American College of Rheumatology Subcommittee on Osteoarthritis Guidelines. Arthritis Rheum. 2000 Sep;43(9):1905-15. doi: 10.1002/1529-0131(200009)43:93.0.CO;2-P. No abstract available. PMID 11014340
- [Background] Drouin JM, Valovich-mcLeod TC, Shultz SJ, Gansneder BM, Perrin DH. Reliability and validity of the Biodex system 3 pro isokinetic dynamometer velocity, torque and position measurements. Eur J Appl Physiol. 2004 Jan;91(1):22-9. doi: 10.1007/s00421-003-0933-0. Epub 2003 Sep 24. PMID 14508689
- [Background] Galan-Mercant A, Baron-Lopez FJ, Labajos-Manzanares MT, Cuesta-Vargas AI. Reliability and criterion-related validity with a smartphone used in timed-up-and-go test. Biomed Eng Online. 2014 Dec 2;13:156. doi: 10.1186/1475-925X-13-156. PMID 25440533
- [Background] Goble DJ. Proprioceptive acuity assessment via joint position matching: from basic science to general practice. Phys Ther. 2010 Aug;90(8):1176-84. doi: 10.2522/ptj.20090399. Epub 2010 Jun 3. PMID 20522675
- [Background] Grob KR, Kuster MS, Higgins SA, Lloyd DG, Yata H. Lack of correlation between different measurements of proprioception in the knee. J Bone Joint Surg Br. 2002 May;84(4):614-8. doi: 10.1302/0301-620x.84b4.11241. PMID 12043789
- [Background] Han J, Waddington G, Adams R, Anson J, Liu Y. Assessing proprioception: A critical review of methods. J Sport Health Sci. 2016 Mar;5(1):80-90. doi: 10.1016/j.jshs.2014.10.004. Epub 2015 Feb 3. PMID 30356896
- [Background] Ho-Pham LT, Lai TQ, Mai LD, Doan MC, Pham HN, Nguyen TV. Prevalence of radiographic osteoarthritis of the knee and its relationship to self-reported pain. PLoS One. 2014 Apr 10;9(4):e94563. doi: 10.1371/journal.pone.0094563. eCollection 2014. PMID 24722559
- [Background] Hurkmans EJ, van der Esch M, Ostelo RW, Knol D, Dekker J, Steultjens MP. Reproducibility of the measurement of knee joint proprioception in patients with osteoarthritis of the knee. Arthritis Rheum. 2007 Dec 15;57(8):1398-403. doi: 10.1002/art.23082. PMID 18050179
- [Background] Jenny JY, Bureggah A, Diesinger Y. Measurement of the knee flexion angle with smartphone applications: Which technology is better? Knee Surg Sports Traumatol Arthrosc. 2016 Sep;24(9):2874-2877. doi: 10.1007/s00167-015-3537-4. Epub 2015 Feb 15. PMID 25682165
- [Background] Kaminski TW, Hartsell HD. Factors Contributing to Chronic Ankle Instability: A Strength Perspective. J Athl Train. 2002 Dec;37(4):394-405. PMID 12937561
- [Background] Kimberlin CL, Winterstein AG. Validity and reliability of measurement instruments used in research. Am J Health Syst Pharm. 2008 Dec 1;65(23):2276-84. doi: 10.2146/ajhp070364. PMID 19020196
- [Background] Knoop J, Steultjens MP, van der Leeden M, van der Esch M, Thorstensson CA, Roorda LD, Lems WF, Dekker J. Proprioception in knee osteoarthritis: a narrative review. Osteoarthritis Cartilage. 2011 Apr;19(4):381-8. doi: 10.1016/j.joca.2011.01.003. Epub 2011 Jan 18. PMID 21251988
- [Background] Kramer J, Handfield T, Kiefer G, Forwell L, Birmingham T. Comparisons of weight-bearing and non-weight-bearing tests of knee proprioception performed by patients with patello-femoral pain syndrome and asymptomatic individuals. Clin J Sport Med. 1997 Apr;7(2):113-8. doi: 10.1097/00042752-199704000-00007. PMID 9113427
- [Background] Kujala UM, Kettunen J, Paananen H, Aalto T, Battie MC, Impivaara O, Videman T, Sarna S. Knee osteoarthritis in former runners, soccer players, weight lifters, and shooters. Arthritis Rheum. 1995 Apr;38(4):539-46. doi: 10.1002/art.1780380413. PMID 7718008
- [Background] Lee D, Han S. Validation of Joint Position Sense of Dorsi-Plantar Flexion of Ankle Measurements Using a Smartphone. Healthc Inform Res. 2017 Jul;23(3):183-188. doi: 10.4258/hir.2017.23.3.183. Epub 2017 Jul 31. PMID 28875053
- [Background] Levinger P, Nagano H, Downie C, Hayes A, Sanders KM, Cicuttini F, Begg R. Biomechanical balance response during induced falls under dual task conditions in people with knee osteoarthritis. Gait Posture. 2016 Jul;48:106-112. doi: 10.1016/j.gaitpost.2016.04.031. Epub 2016 May 6. PMID 27239773
- [Background] Litwic A, Edwards MH, Dennison EM, Cooper C. Epidemiology and burden of osteoarthritis. Br Med Bull. 2013;105:185-99. doi: 10.1093/bmb/lds038. Epub 2013 Jan 20. PMID 23337796
- [Background] Lonn J, Crenshaw AG, Djupsjobacka M, Johansson H. Reliability of position sense testing assessed with a fully automated system. Clin Physiol. 2000 Jan;20(1):30-7. doi: 10.1046/j.1365-2281.2000.00218.x. PMID 10651789
- [Background] Mahmoudian A, van Dieen JH, Baert IA, Jonkers I, Bruijn SM, Luyten FP, Faber GS, Verschueren SM. Changes in proprioceptive weighting during quiet standing in women with early and established knee osteoarthritis compared to healthy controls. Gait Posture. 2016 Feb;44:184-8. doi: 10.1016/j.gaitpost.2015.12.010. Epub 2015 Dec 14. PMID 27004655
- [Background] Marks R. Further evidence of impaired position sense in knee osteoarthritis. Physiother Res Int. 1996;1(2):127-36. doi: 10.1002/pri.6120010208. PMID 9238729
- [Background] Marks R, Quinney HA. Effect of fatiguing maximal isokinetic quadriceps contractions on ability to estimate knee-position. Percept Mot Skills. 1993 Dec;77(3 Pt 2):1195-202. doi: 10.2466/pms.1993.77.3f.1195. PMID 8170768
- [Background] Mourcou Q, Fleury A, Diot B, Franco C, Vuillerme N. Mobile Phone-Based Joint Angle Measurement for Functional Assessment and Rehabilitation of Proprioception. Biomed Res Int. 2015;2015:328142. doi: 10.1155/2015/328142. Epub 2015 Oct 25. PMID 26583101
- [Background] Mourcou Q, Fleury A, Diot B, Vuillerme N. iProprio: a smartphone-based system to measure and improve proprioceptive function. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:2622-2625. doi: 10.1109/EMBC.2016.7591268. PMID 28268860
- [Background] Neogi T, Zhang Y. Epidemiology of osteoarthritis. Rheum Dis Clin North Am. 2013 Feb;39(1):1-19. doi: 10.1016/j.rdc.2012.10.004. Epub 2012 Nov 10. PMID 23312408
- [Background] Nguyen US, Zhang Y, Zhu Y, Niu J, Zhang B, Felson DT. Increasing prevalence of knee pain and symptomatic knee osteoarthritis: survey and cohort data. Ann Intern Med. 2011 Dec 6;155(11):725-32. doi: 10.7326/0003-4819-155-11-201112060-00004. PMID 22147711
- [Background] Nishiguchi S, Yamada M, Nagai K, Mori S, Kajiwara Y, Sonoda T, Yoshimura K, Yoshitomi H, Ito H, Okamoto K, Ito T, Muto S, Ishihara T, Aoyama T. Reliability and validity of gait analysis by android-based smartphone. Telemed J E Health. 2012 May;18(4):292-6. doi: 10.1089/tmj.2011.0132. Epub 2012 Mar 8. PMID 22400972
- [Background] Ockendon M, Gilbert RE. Validation of a novel smartphone accelerometer-based knee goniometer. J Knee Surg. 2012 Sep;25(4):341-5. doi: 10.1055/s-0031-1299669. PMID 23150162
- [Background] Oliveria SA, Felson DT, Reed JI, Cirillo PA, Walker AM. Incidence of symptomatic hand, hip, and knee osteoarthritis among patients in a health maintenance organization. Arthritis Rheum. 1995 Aug;38(8):1134-41. doi: 10.1002/art.1780380817. PMID 7639811
- [Background] Oxford dictionary, accessed on April 19, 2018, https://en.oxforddictionaries.com/definition/smartphone).
- [Background] Ozdalga E, Ozdalga A, Ahuja N. The smartphone in medicine: a review of current and potential use among physicians and students. J Med Internet Res. 2012 Sep 27;14(5):e128. doi: 10.2196/jmir.1994. PMID 23017375
- [Background] Paillard, J., & Brouchon, M. (1968). Active and passive movements in the calibration of position sense. The neuropsychology of spatially oriented behavior. In: S.J. Freedman (ed), The neuropsychology of spatially oriented behavior, Dorsey Press, Homewood III., chap. 3, 37-55.
- [Background] Piriyaprasarth P, Morris ME, Winter A, Bialocerkowski AE. The reliability of knee joint position testing using electrogoniometry. BMC Musculoskelet Disord. 2008 Jan 22;9:6. doi: 10.1186/1471-2474-9-6. PMID 18211714
- [Background] Pourahmadi MR, Ebrahimi Takamjani I, Sarrafzadeh J, Bahramian M, Mohseni-Bandpei MA, Rajabzadeh F, Taghipour M. Reliability and concurrent validity of a new iPhone(R) goniometric application for measuring active wrist range of motion: a cross-sectional study in asymptomatic subjects. J Anat. 2017 Mar;230(3):484-495. doi: 10.1111/joa.12568. Epub 2016 Dec 2. PMID 27910103
- [Background] Pourahmadi MR, Taghipour M, Jannati E, Mohseni-Bandpei MA, Ebrahimi Takamjani I, Rajabzadeh F. Reliability and validity of an iPhone((R)) application for the measurement of lumbar spine flexion and extension range of motion. PeerJ. 2016 Aug 23;4:e2355. doi: 10.7717/peerj.2355. eCollection 2016. PMID 27635328
- [Background] Relph N, Herrington L. Criterion-related validity of knee joint-position-sense measurement using image capture and isokinetic dynamometry. J Sport Rehabil. 2015 Jan 13;24(1):2013-0119. doi: 10.1123/jsr.2013-0119. Print 2015 Feb 1. PMID 25310567
- [Background] Romero-Franco N, Montano-Munuera JA, Jimenez-Reyes P. Validity and Reliability of a Digital Inclinometer to Assess Knee Joint-Position Sense in a Closed Kinetic Chain. J Sport Rehabil. 2017 Jan;26(1):jsr.2015-0138. doi: 10.1123/jsr.2015-0138. Epub 2016 Aug 24. PMID 27632887
- [Background] S Edwards E, Lin YL, H King J, R Karduna A. Joint position sense - There׳s an app for that. J Biomech. 2016 Oct 3;49(14):3529-3533. doi: 10.1016/j.jbiomech.2016.07.033. Epub 2016 Aug 8. PMID 27567568
- [Background] Smith TO, Davies L, Hing CB. A systematic review to determine the reliability of knee joint position sense assessment measures. Knee. 2013 Jun;20(3):162-9. doi: 10.1016/j.knee.2012.06.010. Epub 2012 Jul 20. PMID 22819143
- [Background] Tsauo JY, Cheng PF, Yang RS. The effects of sensorimotor training on knee proprioception and function for patients with knee osteoarthritis: a preliminary report. Clin Rehabil. 2008 May;22(5):448-57. doi: 10.1177/0269215507084597. PMID 18441041
- [Background] Yoo JJ, Kim DH, Kim HA. Risk factors for progression of radiographic knee osteoarthritis in elderly community residents in Korea. BMC Musculoskelet Disord. 2018 Mar 12;19(1):80. doi: 10.1186/s12891-018-1999-5. PMID 29530005
- [Background] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Background] Zhu R, Zhou Z. A real-time articulated human motion tracking using tri-axis inertial/magnetic sensors package. IEEE Trans Neural Syst Rehabil Eng. 2004 Jun;12(2):295-302. doi: 10.1109/TNSRE.2004.827825. PMID 15218943
- [Result] Ferretti A, Valeo L, Mazza D, Muliere L, Iorio P, Giovannetti G, Conteduca F, Iorio R. Smartphone versus knee ligament arthrometer when size does not matter. Int Orthop. 2014 Oct;38(10):2197-9. doi: 10.1007/s00264-014-2432-9. Epub 2014 Jul 9. PMID 25005461